CLINICAL TRIAL: NCT05951101
Title: Evaluation of the Safety and Performance of the Zenith LAA Occlusion System and Procedure for the Mechanical Closure of the Left Atrial Appendage (LAA)
Brief Title: Zenith LAA Occlusion System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AuriGen Medical Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CLN002
Record Dates: First submitted 2023-06-29; First posted 2023-07-18 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Atrial Fibrillation; Left Atrial Appendage; Stroke
Keywords: LAA Occlusion; Left Atrial Appendage; Atrial Fibrillation; LAA closure
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Intervention Model Description: Implantation of Zenith LAA Occlusion System
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Zenith LAA Occlusion System (Experimental): Zenith LAA Occlusion System Implantation
  Interventions: Device: Zenith LAA Occlusion System

INTERVENTIONS:
Device: Zenith LAA Occlusion System — LAA closure in patients with non-valvular atrial fibrillation, with an ostial diameter between 17 mm and 25 mm

SUMMARY:
Demonstrate the safety and performance of the Zenith LAA Occlusion System and procedure to occlude the Left Atrial Appendage (LAA) from the left atrium (LA) using a minimally invasive technique.

Indication - LAA closure in patients with non-valvular atrial fibrillation, with an ostial diameter between 18 mm and 26 mm

DETAILED DESCRIPTION:
The study objective is to demonstrate the safety and performance of the Zenith LAA Occlusion System and procedure to occlude the Left Atrial Appendage (LAA) from the left atrium (LA) using a minimally invasive technique.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 at the time of screening
2. Documented diagnosis of non-valvular AF
3. Clinical indication for LAA occlusion
4. Willing and able to return to and comply with scheduled follow-up visits and testing, including medical treatment as required by the protocol.
5. Willing and able to provide written informed consent

Exclusion Criteria:

Within 30 days before the procedure date:

1. Exhibited NYHA class III or IV heart failure symptoms
2. Known bleeding disorders (such as bleeding diathesis, thrombocytopenia [platelet count <100 X 109/L], severe anaemia [haemoglobin of <8 g/dL], or INR >2 [spontaneous])

   Within 90 days before the procedure date:
3. Documented history of myocardial infarction or unstable angina
4. Documented embolic stroke, TIA or suspected neurologic event
5. Chronic renal insufficiency (eGFR ≤15mL/min per 1.73 m2 (CKD-EPI)) or end-stage renal disease
6. Requires long-term oral anticoagulation therapy for a condition other than AF
7. Diagnosed active local or systemic infection, septicaemia, active pericarditis, or fever of unknown origin
8. Known acquired or inherited propensity for forming blood clots (e.g., malignancy and factor V Leiden mutation) established by prior objective testing
9. Contraindication to the standard of care post-implantation antithrombotic medication regime (e.g., dual antiplatelet therapy (DAPT)/direct oral anticoagulant (DOAC)
10. Rheumatic heart disease
11. Implanted mechanical valve prosthesis
12. Documented carotid disease, defined as greater than 70% stenosis without symptoms or greater than 50% stenosis with symptoms
13. Body mass index greater than 40 kg/m2
14. Patient is pregnant or breastfeeding or plans/desires to get pregnant within the next 12 months post-procedure
15. Current or planned enrolment in an investigation or study of an investigational device or investigational drug that would interfere with this study and the required follow-up
16. Mental impairment or other psychiatric conditions which may not allow the patient to understand the nature, significance, and scope of the study
17. Any other criteria (including physical and mental health), medical illness, or comorbidity which would make the subject unsuitable to participate in this study as determined by the clinical site principal investigator
18. Patients with known allergy or sensitivity to nitinol (nickel and titanium) or any of the other materials in the Zenith LAA Occlusion System Implant
19. Life expectancy of less than 1 year
20. Inability, unwillingness, or contraindication to undergo Trans-Oesophageal and/or Trans-Thoracic Echocardiogram (TOE/TTE) or Cardiac Computed Tomography Angiography (CCTA) imaging or any catheterisation procedures
21. Any anatomical condition that precludes the patient from undergoing LAA occlusion with the AuriGen Zenith LAA Occlusion System implant procedure, as determined by the principal investigator

    Imaging Exclusion Criteria:
22. Patients with a maximal ostial left atrial appendage diameter >25 mm or <17 mm by pre-procedural ECG-gated CT scan, to fit the Zenith LAA Occlusion System
23. Patients where CCTA analysis suggests that the Zenith LAA Occlusion System may not be suitable
24. Intracardiac thrombus diagnosed by CCTA or echocardiography
25. Previous occlusion/ligation of the LAA (by any surgical or percutaneous method)
26. Documented presence of implanted closure devices (e.g. Atrial septal defect (ASD), Patent foramen ovale (PFO) or Ventricular septal defect (VSD) device) for congenital defect treatment
27. Documented Left Ventricular Ejection Fraction (LVEF) <30%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Procedural success | 72 hours
  Acute procedural success is defined as the delivery and release of the Zenith LAA Occlusion System in the target location (LAA) without any device or procedure related serious adverse events until the post-procedure discharge or 72 hours (whichever comes first)
Mechanical device closure | 45 days
  Mechanical device closure - residual jet around the device ≤5 mm at 45 days by TOE

SECONDARY OUTCOMES:
Device related thrombus | 45 days and 12 months
  LAAO device-related thrombus as assessed by TOE at 45 days and by CCTA at 12 months
SAE | through study completion, an average of 1 year
  All SAEs device and/or procedure-related post-procedure and to the end of the study
Stroke | 12 months
  Ischemic stroke through 12 months
Thromboembolism | 12 months
  Systemic thromboembolism through 12 months
Device closure | 6 months
  Mechanical device closure - residual jet around the device ≤5 mm at 6 months (if it is not achieved at 45 Days)
Device use questionnaire | up to 24 hours
  Use of the Zenith LAA Occlusion System per Device use questionnaire (Operator)
Changes in Quality of Life score according to SF-12 questionnaire | Baseline, 45 days, 6 months and 12 months
  Patient-reported health quality at Baseline, 45 days, 6 months, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Felix Mahfoud, Principal Investigator — Internal Medicine and Cardiology, Saarland University Hospital; Christian Ukena, Principal Investigator — Saarland University Hospital; Sandeep Panikker, Principal Investigator — University Hospitals Coventry & Warwickshire NHS Trust
Locations (3):
- The Royal Melbourne Hospital, Parkville, Victoria, Australia
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch

IPD SHARING:
Plan to Share IPD: No